CLINICAL TRIAL: NCT06892483
Title: Breastmilk Composition in Response to a Bout of Exercise
Brief Title: Breastmilk in Response to a Bout of Exercise
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Pataky, Principal Investigator, Mayo Clinic
Other Study IDs: 24-006207
Record Dates: First submitted 2025-03-13; First posted 2025-03-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Infant Development; Obesity, Childhood; Diabetes, Childhood-Onset
Keywords: Breast milk; Postpartum exercise
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus | interventions — Total Quality Management; Adiposity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Blood samples and breastmilk will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active: Exercise > 3 days per week of moderate-intensity exercise
  Interventions: Other: Pre-Pregnancy BMI
- Inactive: ≤ 1 day per week of exercise
  Interventions: Other: Pre-Pregnancy BMI

INTERVENTIONS:
Other: Pre-Pregnancy BMI — Pre-pregnancy BMI between 18.5-24.99
  Other Names: Lean
Other: Pre-Pregnancy BMI — Pre-pregnancy BMI between 25-39.99
  Other Names: Obese

SUMMARY:
The purpose of this study is to unveil the mechanistic benefits of a bout of postpartum maternal exercise on infant health that are provided by breastmilk.

DETAILED DESCRIPTION:
The nutrients and antibodies in breastmilk promote infant growth, development, and immunity. Breastfed infants exhibit lower risk of adult-onset obesity and type 2 diabetes compared to formula-fed infants, and the composition of breastmilk is influenced by maternal factors such as obesity and type 2 diabetes, profoundly impacting its health benefits. While postpartum maternal exercise enhances infant health, its effects on breastmilk composition remain unknown, hindering our understanding of how postpartum exercise benefits breastfed infants.

ELIGIBILITY:
Exclusion Criteria:

* Active coronary artery disease or heart failure.
* Participation in a structured exercise program ≥ 1 day/week in the "inactive" subcohort or < 3 days per week in the "active" subcohort.
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  * Abnormal liver function test results (Transaminase >2 times the upper limit of normal
  * Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2);
  * If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
  * Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L); testing required within three months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
  * Abuse of alcohol or recreational drugs
  * Active tobacco smoking within the past 3 months
  * Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis).
  * Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg) at the time of screening.
  * A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
  * Active pregnancy
  * Restrictions on Use of Other Drugs or Treatments:

    * Any other medication believed to be a contraindication to the subject's participation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Lactating Females
Study Population: Depending upon mode of delivery, it may take up to 6-8 weeks to return to pre-pregnancy physical activity levels, and participants may prefer to have their postpartum visit to receive "medical clearance". Thus, by 2 months after delivery, most participants will have been medically cleared to exercise. Recruitment and screening of participants will take primarily place in the clinical setting either prior to or within 2 months of giving birth. Participants will be consulted throughout the >2-month period postpartum by an Internationally Board-Certified Lactation Consultant on the study team to increase the likelihood of successful breastfeeding for participants that are recruited prior to giving birth. Half of the participants will be enrolled with a pre-pregnancy BMI between 18.5-24.99 (n=30; normal weight) and the other half will be between 25-39.99 (n=30; obese). The participant's first recorded first-trimester BMI will be used.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-10-10 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Breastmilk Exosome Concentration | 1 month
  The molecules in small extracellular vesicles (exosomes) can transmit information between cells throughout the body. A bout of exercise induces a robust release of exosomes in the plasma with unique molecular cargo. Exosomes are also present in breastmilk, and there is evidence that breastmilk exosomes can evade degradation in the infant gut and can thus transmit molecular information from mother to infant. Though maternal exercise is viewed as beneficial for the breastfeeding infant, the molecular mechanisms of how this occurs remain unknown. The primary objective of this trial will be to determine if a bout of maternal exercise increases the release exosomes in breastmilk. The investigators will measure breastmilk exosome concentration using nano particle tracking.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pataky, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided